CLINICAL TRIAL: NCT02917161
Title: Prostatic Artery Embolization Before Radical Prostatectomy in Prostate Cancer: A Proof-of-concept Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dominik Abt (Other)
Responsible Party: Sponsor-Investigator, Dominik Abt, Dr. med., Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTU 15/015
Record Dates: First submitted 2016-09-24; First posted 2016-09-28 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: Prostate; Prostatic Neoplams; Therapeutic Embolization; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prostatic Artery Embolization (PAE) (Experimental): PAE is performed 6weeks before RALP
  Interventions: Device: Prostatic Artery Embolization (PAE)

INTERVENTIONS:
Device: Prostatic Artery Embolization (PAE) — PAE is performed 6 weeks before radical prostatectomy

SUMMARY:
MRI findings after successful PAE in patients suffering from BPH suggest a complete necrosis of the prostate after this intervention. Thus, PAE might also play a role in the treatment of prostate cancer.

This proof of concept study assess the impact of PAE in patients with proven prostate cancer.

DETAILED DESCRIPTION:
MRI findings after successful PAE in patients suffering from BPH suggest a complete necrosis of the prostate after this intervention. Thus, PAE might also play a role in the treatment of prostate cancer.

This proof of concept study assess the impact of PAE in patients with proven prostate cancer.

PAE is performed in patients that are planned to undergo robot-assisted laparoscopic prostatectomy for proven localized prostate cancer.

The impact of neo-adjuvantly performed PAE on histological tumor regression, surgical margins as well as on safety parameters are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men 45 - 75 years old undergoing RALP
* Patient has biopsy-proven prostate adenocarcinoma
* Localized disease (tumorstage cT1-cT2), assessed by clinical and MRI findings
* Written informed consent

Exclusion Criteria:

* Severe atherosclerosis
* Severe tortuosity or ectasia in the aortic bifurcation or internal iliac arteries
* Tumor stage > cT2 assessed by clinical and MRI findings
* Allergy to intravenous contrast media
* Contraindication for MRI imaging
* Renal failure (GFR<60ml/min)
* History of pelvic irradiation or radical pelvic surgery

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09; Primary Completion 2017-06 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Tumor response | 6 weeks after PAE (at the time of RALP)
  Histological assessment of the excised prostate to determine whether pathological complete response was achieved, defined as complete absence of histologically identifiable cancer cells in the excised prostate.

SECONDARY OUTCOMES:
Histological Tumor Regression Grade | 6 weeks after PAE (at the time of RALP)
Surgical margins assessment (R0 /R1) | 6 weeks after PAE (at the time of RALP)
  - Success of radical prostatectomy defined as the complete resection of cancerous prostate gland tissue and completely negative surgical margins.
Assessment of Adverse Events of PAE according to CTCAE V4.03 | At the time of PAE and 6 weeks afterwards
Assessment of Adverse Events of PAE according to Clavien-Dindo classification | At the time of PAE and 6 weeks afterwards
Assessment of Adverse Events of RALP after PAE according to CTCAE V4.03 | At the time of RALP, 6 weeks and 12 weeks later
Assessment of Adverse Events of RALP after PAE according to Clavien-Dindo classification | At the time of RALP, 6 weeks and 12 weeks later
Change of prostate volume in MRI after PAE | Before and 6 weeks after PAE
Change of tumor detection rate in MRI after PAE | Before and 6 weeks after PAE
Change of tumor size in MRI after PAE | Before and 6 weeks after PAE
Change of PIRADS classification in MRI after PAE | Before and 6 weeks after PAE

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Abt, MD, Principal Investigator — Cantonal Hospital of St. Gallen; Livio Mordasini, MD, Principal Investigator — Cantonal Hospital Luzerne
Locations (2):
- Switzerland (2):
  - Cantonal Hospital Lucerne, Department of Urology, Lucerne
  - Urological Department, Cantonal Hospital of St. Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No